CLINICAL TRIAL: NCT01018953
Title: Phase II, Open, Adaptive, Dose Escalating, Multicentre Titration Study to Assess the Efficacy and Safety of Repeated Subcutaneous Administration of Different Doses of BIM 23A760 in Patients With Carcinoid Syndrome
Brief Title: Study to Assess the Efficacy and Safety of Different Doses of BIM 23A760 in Patients With Carcinoid Syndrome
Acronym: CAMPANULA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary data from study NCT00994214 do not support expected inhibition of GH and IGF-1
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8-55-52060-004; 2009-013222-16 (EudraCT Number)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Carcinoid Syndrome
MeSH Terms: conditions — Serotonin Syndrome | interventions — TBR-760

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIM 23A760 (Experimental): This dose adaptive study is planned to treat up to 20 patients in each starting dose cohort, with a maximum of three starting dose cohorts. The doses planned to be assessed are 1, 2, 4, 6 and 8 mg, however, the maximum starting dose will be 4 mg. The starting dose of the first cohort will be 1 mg; the first cohort will include at least five patients. After the first fifteen patients have been treated for 4 weeks, the results will be reviewed by a Data Review Committee. An extension phase (Part B) is planned for those subjects completing the initial study and fulfilling specific eligibility criteria (symptoms control, willingness to participate, safety and tolerability).
  Interventions: Drug: BIM 23A760

INTERVENTIONS:
Drug: BIM 23A760 — BIM 23A760 is a solution at a concentration of 5 mg/mL ready for subcutaneous injection. BIM 23A760 dose of 1, 2, 4, 6 and 8 mg can be given to the patient according to a dose escalation and titration process. Patients will receive 24 weekly injections of BIM 23A760 during the treatment period. Patients eligible to continue the extension phase will be administered BIM 23A760 for further 52 weekly injections.

SUMMARY:
The purpose of the protocol is to assess the efficacy and safety of BIM 23A760 on patient's overall satisfaction in terms of symptom relief (diarrhoea and/or flushes) in patients with carcinoid syndrome after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a carcinoid syndrome defined as ≥3 stools/day and/or ≥3 flushes/week.
* The patient has elevated 5-Hydroxyindoleacetic acid (above upper limit normal).
* The patient has a well-differentiated mid-gut carcinoid tumour or serotonin secreting tumour of unknown localisation with hepatic metastasis.

Exclusion Criteria:

* The patient has undergone surgery related to a neuroendocrine tumour (NET) within 4 weeks prior to study entry or has surgery planned during the study.
* The patient has received short acting somatostatin analogues (SSAs) within 2 weeks before study entry or has received short acting SSAs for more than 3 months.
* The patient has received a radiolabelled SSA at any time before study entry.
* The patient has received long acting SSAs under certain circumstances.
* The patient has previously received any specific anti tumour treatment such as chemotherapy, (chemo)embolisation, radiotherapy or interferon in the last 6 months.
* The patient has signs or symptoms of cardiac insufficiency.
* The patient has an ejection fraction <40% and/or clinically severe cardiac valvular regurgitation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (54):
- University Hospital, Internal Medicine - Oncology, Vienna, Austria
- Belgium (3):
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - UZ GAsthuisberg, Leuven
- Czechia (3):
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultní nemocnice Na Bulovce, Ústav radiační onkologie, Prague
- Finland (2):
  - Helsinki Central University Hospital, Helsinki
  - Turku University Hospital, Turku
- France (5):
  - Service de Gastroentérologie, Clichy
  - Unité d'Oncologie Médicale, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre René Gauducheau, Nantes
  - Unité de Gastro-Entérologie, Villejuif
- Germany (3):
  - Charite Universitätsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mainz, Mainz
- St James's Hospital, Dublin, Ireland
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (6):
  - Università degli Studi di Bologna, Policlinico S. Orsola-Malpighi, Bologna
  - Istituti Ospitalieri di Cremona, Cremona
  - Ospedale San Martino, Genova
  - AO Universitaria Policlinico di Modena, Modena
  - Ospedale S.Maria della Misericordia, Perugia
  - Università degli Studi di Roma "La Sapienza", II Facoltà di Medicina e Chirurgia, Ospedale Sant'Andrea, Roma
- Latvia (2):
  - Latvian Oncology centre of Riga Eastern Clinical University Hospital, Riga
  - Vidzemes Hospital, Valmiera
- Netherlands (2):
  - UMCG, Groningen
  - Erasmus MC, Rotterdam
- Poland (4):
  - Centrum Onkologii Instytut im.M. Sklodowskiej-Curie oddzial w Gliwicach, Gliwice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Instytut im Marii Sklodowskiej Curie, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Wroclaw, 50-367
- Russia (7):
  - Altay Regional Oncology dispensary, Barnaul
  - Republican Clinical Oncology dispensary of the Ministry of Health of Republic of Tatarstan, Kazan'
  - Non-state Institution of Public health "Central Clinical hospital # 1, public corporation "Russian railways", Moscow
  - St-Petersburg State Medical University named after academician Pavlov I.P., Saint Petersburg
  - St-Petersburg State Institution of Public Health City Clinical Oncology dispensary, Saint Petersburg
  - Tula Regional Oncology Dispensary, Tula
  - Voronezh Regional Clinical Oncology Dispensary, Voronezh
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - Martinska fakultna nemocnice, Martin
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Son Dureta, Palma de Mallorca
- Akademiska Hospital, Dept of Oncology & Endocrinology, Uppsala, Sweden
- Ukraine (2):
  - Donetsk National Medical University named after M. Gorkiy, Donetsk Regional Antitumor Center, Donetsk
  - Uzhgorod national university, Postgraduate faculty, Uzhgorod Central City Clinical Hospital, Uzhhorod
- United Kingdom (5):
  - University Hospital Aintree, Liverpool
  - St Bartholomew's Hospital, London
  - Royal Free Hospital, London
  - Christie Hospital and Holt Radium Institute, Manchester
  - Royal Preston Hospital, Sharoe Green Lane, Lancashire, Preston

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated prematurely. Only 8 patients were treated in part A and no patients participated in part B.
Pre-assignment Details: Patients screened were 15 and not treated were 7 (2 subjects were not included due to early termination of study by sponsor and 5 subjects failed to meet inclusion criteria).
Groups:
- BIM 23A760: This dose adaptive study was planned to treat up to 20 patients in each starting dose cohort, with a maximum of three starting dose cohorts. The doses planned to be assessed were 1, 2, 4, 6 and 8 mg; however, the maximum starting dose was 4 mg. The starting dose of the first cohort was 1 mg and the first cohort would include at least five patients. After the first 15 patients were treated for 4 weeks, the results were to be reviewed by a Data Review Committee. An extension phase (Part B) was planned for those subjects completing the initial study and fulfilling specific eligibility criteria (symptoms control, willingness to participate, safety and tolerability).
  BIM 23A760 was a solution at a concentration of 5 mg/mL ready for subcutaneous injection. BIM 23A760 doses of 1, 2, 4, 6 and 8 mg were to be given to the patient according to a dose escalation and titration process. Patients would have received 24 weekly injections of BIM 23A760 during the treatment period.
Period: Overall Study
Arm/Group | BIM 23A760
Started | 8
BIM 23A760 1 mg | 3
BIM 23A760 2 mg | 2
BIM 23A760 4 mg | 3
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Study termination by sponsor | 5

BASELINE CHARACTERISTICS:
Arm/Group | BIM 23A760
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (6.88)
Age, Customized [Number; unit: participants]
  Between 18 and 75 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/ White | 8
Region of Enrollment [Number; unit: participants]
  Russian Federation | 1
  United Kingdom | 2
  Netherlands | 1
  Belgium | 1
  Ireland | 1
  Finland | 1
  Germany | 1
Diabetic status [Number; unit: participants]
  Diabetic | 0
  Nondiabetic | 8
Post-menopausal status [Number; unit: participants]
  Yes | 6
  No | 0
  N/A - Not applicable | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Positive Overall Satisfactory Relief of Symptoms (Diarrhoea and/or Flushes) on the Likert Scale
Description: Patient satisfaction based on a Likert scale from 0-5 (0 being not satisfied and 5 being completely satisfied)
Time Frame: Week 24
Population: Study was prematurely terminated and no data was collected/analyzed for this outcome measure.
Arm/Group | BIM 23A760
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Patients With Improvement in Symptoms (Diarrhoea and/or Flushes)
Time Frame: Up to week 24
Population: Study was prematurely terminated and no data was collected/analyzed for this outcome measure.
Arm/Group | BIM 23A760
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in the Quality of Life (QoL) Assessment
Time Frame: Week 24
Population: Study was prematurely terminated and no data was collected/analyzed for this outcome measure.
Arm/Group | BIM 23A760
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in 5 Hydroxyindoleacetic Acid (5 HIAA) and Chromogranin A
Time Frame: Week 24
Population: Study was prematurely terminated and no data was collected/analyzed for this outcome measure.
Arm/Group | BIM 23A760
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Subjects Reported Adverse Events, Including Any Findings From an Examination of the Injection Site(s)
Time Frame: Up to week 26
Population: Both ITT (Intent-To-Treat) and safety populations were the same analysis group. Treatment emergent adverse events (TEAE) reported by 2 or more patients (safety population) by primary system organ class.
Measure: Number; unit: Participants
Arm/Group | BIM 23A760
Number analyzed (Participants) | 8
Participants
  General Disorders & Administration Site Condition | 5
  Gastrointestinal Disorder | 4
  Nervous System Disorders | 3
  Infections and Infestations | 2
  Metabolism and Nutritional Disorders | 2
  Neoplasms Benign, Malignant and unspecified | 2
  Reproductive System and Breast Disorders | 2

6. Secondary Outcome: Minimum Concentration (Cmin) BIM 23A760 Plasma Levels
Time Frame: At 9 timepoints up to 1 week after 24th administration in week 24
Population: Study was prematurely terminated and no data was collected/analyzed for this outcome measure.
Arm/Group | BIM 23A760
Number analyzed (Participants) | 0

7. Secondary Outcome: Concentration at 2 Hours Postdose (C2 Hours) BIM 23A760 Plasma Levels
Time Frame: At 8 timepoints up to week 24
Population: Study was prematurely terminated and no data was collected/analyzed for this outcome measure.
Arm/Group | BIM 23A760
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to week 26
Description: Dose received prior to AE onset.
  Two serious adverse events (SAEs) 'Confusional State' and 'Nausea' were not included as they occurred during screening phase, before starting study drug.
Arm/Group | BIM 23A760
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIM 23A760 (N=8)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIM 23A760 (N=8)
Injection site erythema (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Injection site inflammation (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (3)
Injection site pruritus (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucous stools (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peripheral vascular system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to premature termination of the study, no data was collected/analyzed and no patient participated in Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No